CLINICAL TRIAL: NCT07092787
Title: Reducing Smartphone Overuse for Adolescents With Attention-Deficit Hyperactive Disorder: A Randomized Controlled Trial
Brief Title: Reducing Smartphone Overuse for Adolescents With Attention-Deficit Hyperactive Disorder
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Education University of Hong Kong (Other)
Responsible Party: Principal Investigator, YUM Yen Na Cherry, Associate Professor, Education University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2023-2024-0412; HHB/H/41/208 (Other Grant/Funding Number: Health Bureau, Hong Kong SAR)
Record Dates: First submitted 2025-07-10; First posted 2025-07-30 (Actual); Last update posted 2025-07-30 (Actual); Status verified 2025-07

CONDITIONS: Attention Deficit Hyerpactivity Disorder; Smartphone Addiction
MeSH Terms: conditions — Internet Addiction Disorder

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Smartphone Intervention (Experimental): The treatment group will receive a 12-week individualized smartphone-based behavioral intervention based on the following strategies. They will be contacted once a week to collect the objective smartphone use patterns and check for compliance of the intervention strategies.
  Interventions: Behavioral: Smartphone-based behavioral intervention
- Control (Placebo Comparator): The control group will receive information about the known benefits and risks of SO and activate their smartphones' screentime monitoring setting. They will be contacted once a week to collect the objective smartphone use patterns, but they will self-monitor their smartphone usage.
  Interventions: Other: Self-monitoring of smartphone use

INTERVENTIONS:
Behavioral: Smartphone-based behavioral intervention — The proposed study will use a behavioral smartphone-based intervention in a 12-week RCT among clinically diagnosed ADHD adolescents in Hong Kong. Guided by a conceptual framework on SO in ADHD, we will implement specific strategies that counter the potentially addictive qualities of smartphones using built-in smartphone functions that have been previously shown to be effective.
  Arms: Smartphone Intervention
Other: Self-monitoring of smartphone use — Participants will receive information about the known benefits and risks of SO and activate their smartphones' screentime monitoring setting. They will receive weekly reminders to submit their smartphone usage data.
  Arms: Control

SUMMARY:
This study will develop and evaluate a smartphone-based behavioral intervention for adolescents with Attention-Deficit Hyperactive Disorder (ADHD) and smartphone overuse in Hong Kong. The main questions it aims to answer are:

* Can a smartphone-based intervention lower self-reported smartphone dependence and objective smartphone usage?
* Can a smartphone-based intervention lower parent-rated and self-rated ADHD symptoms?
* Are there differences in electroencephalogram (EEG) in the smartphone salient vs smartphone non-salient conditions after intervention?

Adolescent participants will:

* report weekly smartphone use patterns based on app screencap for 12 weeks
* complete online surveys on smartphone dependency and ADHD symptoms for 3 times
* receive 10-minute EEG recordings to gather resting-state EEG data in a natural and relaxing state for 3 times

Parent participants will:

* provide a valid clinical report to confirm the adolescent's diagnosis of ADHD
* complete online surveys to report on the adolescent's smartphone usage and ADHD symptoms for 3 times

ELIGIBILITY:
Inclusion Criteria:

* full-scale IQ above 85
* right-handedness to control for hemispheric dominance
* a confirmed diagnosis of ADHD
* ratings of current symptoms of ADHD on the Strengths and Weaknesses of Attention Deficit Hyperactivity Disorder Symptoms and Normal Behaviour Scale
* on a stable dose of ADHD medication for at least 4 weeks prior to trial entry or was taking no medication, with no plan to start or change medication type or dosage for the duration of the study
* over 2 hours of daily smartphone use within the last 4 weeks excluding educational apps
* a total score on the Smartphone Addiction Scale - Short Version (SAS-SV) above 31 and 33 for male and female adolescents, respectively

Exclusion Criteria:

* severe physical or sensory disabilities that may alter the participation in the intervention
* major depressive episode, bipolar disorder, substance abuse/dependence within the last 6 months
* significant neurological conditions (e.g., epilepsy, traumatic brain injury) that could affect cognitive and behavioral functioning
* concurrent participation in other ADHD interventions (e.g., clinical trials) excluding standard care

Ages: 12 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 120 (Estimated)
Dates: Start 2025-09 (Estimated); Primary Completion 2028-03 (Estimated); Study Completion 2028-06 (Estimated)

PRIMARY OUTCOMES:
Minutes of smartphone use | Baseline, 1, 2, 3, 4, 5, 6, 7, 8, 9, 10, 11, 12, 13 weeks, and 12 months
  Objective smartphone use data will be collected via smartphone apps (e.g., "ScreenTime" on Apple or "Digital Wellbeing" on Android) to trace the pattern of smartphone use of each participant. Participants will send screenshots of the minutes of smartphone use over the previous 7 days on their phones.
Categories of smartphone use | Baseline, 1, 2, 3, 4, 5, 6, 7, 8, 9, 10, 11, 12, 13 weeks, and 12 months
  Objective smartphone use data will be collected via smartphone apps (e.g., "ScreenTime" on Apple or "Digital Wellbeing" on Android) to trace the pattern of smartphone use of each participant. Participants will send screenshots of the distribution of minutes spent according to categories of use (social networking, games, entertainment, productivity, etc.) over the previous 7 days on their phones.
Number of screen unlocks or "pickups" | Baseline, 1, 2, 3, 4, 5, 6, 7, 8, 9, 10, 11, 12, 13 weeks, and 12 months
  Objective smartphone use data will be collected via smartphone apps (e.g., "ScreenTime" on Apple or "Digital Wellbeing" on Android) to trace the pattern of smartphone use of each participant. Participants will send screenshots of the number of screen unlocks or "pickups" over the previous 7 days on their phones.
Number of notifications | Baseline, 1, 2, 3, 4, 5, 6, 7, 8, 9, 10, 11, 12, 13 weeks, and 12 months
  Objective smartphone use data will be collected via smartphone apps (e.g., "ScreenTime" on Apple or "Digital Wellbeing" on Android) to trace the pattern of smartphone use of each participant. Participants will send screenshots of the number of notifications received over the previous 7 days on their phones.
Smartphone dependence | Baseline, 13 weeks, and 12 months
  To allow for comparisons with existing studies, we will use the Smartphone Addiction Scale - Short Version validated in Hong Kong, which was designed for the assessment of smartphone dependence and showed good reliability and validity. The scale has ten items, such as "Missing planned work due to smartphone use" and "I will never give up using my smartphone even when my daily life is already greatly affected by it". Each item was measured by 6-point scales, from 1= "strongly disagree" to 6 = "strongly agree". Total score on the scale will be used to assess the degree of each participant's smartphone dependence, with suggested cut-off values of smartphone overuse for male and female was 31 and 33, respectively.

SECONDARY OUTCOMES:
ADHD symptoms | Baseline, 13 weeks, and 12 months
  Parents will rate their child's behaviors on a 7-point scale using the Strengths and Weaknesses of Attention Deficit Hyperactivity Disorder Symptoms and Normal Behaviour Scale, which rephrased the 18 ADHD items of the DSM into neutral or positive statements. Scores of each statement range from -3 (far above average) to +3 (far below average), anchoring on normative behavior in age-matched adolescents. Two subscales on inattention and hyperactivity-impulsivity symptoms can be derived. Adolescents will also self-rate their ADHD symptoms.
Resting-state EEG frequency | Baseline, 13 weeks, and 12 months
  During the EEG recording process, adolescent participants will be asked to relax and avoid swallowing and movements that may cause artifacts. For 5 min of recording, participants will look at a blank piece of paper on the table. For another 5 min of recording, they will look at their own smartphone, face-down with notifications and sound turned off, on the table. The order will be counterbalanced across participants. The target outcome measures are alpha (8-12Hz) and delta (1-4Hz) EEG frequency bands.

CONTACTS AND LOCATIONS:
Overall Officials: Yen Na Yum, Principal Investigator — The Education University of Hong Kong

IPD SHARING:
Plan to Share IPD: No
Aggregate and anonymized data will be shared in open access publications, but individual participant data will not shared to protect the privacy of the participants, as stipulated in the ethical review approval.

REFERENCES:
- [Derived] Yum YN, Li X, Poon KY, Leung CH. Reducing smartphone overuse for adolescents with attention-deficit hyperactive disorder: study protocol for a randomized controlled trial. BMC Psychiatry. 2025 Oct 31;25(1):1043. doi: 10.1186/s12888-025-07493-w. PMID 41174591